CLINICAL TRIAL: NCT04649736
Title: Prevalence of Altered Pulmonary Function Post-infection by COVID-19 and Impact of Participation in a Pilot Program of Comprehensive Rehabilitation in the Short and Medium-term
Brief Title: Home-based Respiratory Physiotherapy and Telephone-Based Psychological Support in Severe COVID-19 Patients
Acronym: WAYRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Johns Hopkins University (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202852
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Respiratory Disease; Mental Health Disorder
Keywords: COVID-19; Mental Health; Respiratory Function Tests; Physical and Rehabilitation Medicine; Quality of Life
MeSH Terms: conditions — COVID-19; Respiration Disorders; Mental Disorders; Psychological Well-Being | interventions — Respiratory Rate; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Respiratory Physiotherapy and Telephone-Based Psychological Support (Experimental): Participants in the intervention arm will receive the conventional care given by the hospital that consists of discharged recommendations and a follow-up plan through telephone calls to verify treatment compliance. Discharged recommendations include performing respiratory exercises at home and medication. There is no plan for diagnosing mental illness or a strategy for respiratory o psychological rehabilitation at the hospital.
  Additionally, these participants will receive the intervention program that involves home-based respiratory physiotherapy and telephone-based psychological support for 6 weeks.
  Interventions: Other: Respiratory and psychological rehabilitation
- Control (No Intervention): Participants in the control arm will only receive the conventional care given by the hospital that consists of discharged recommendations and a follow-up plan through telephone calls to verify treatment compliance. Discharged recommendations include performing respiratory exercises at home and medication. There is no plan for diagnosing mental illness or a strategy for respiratory o psychological rehabilitation at the hospital.

INTERVENTIONS:
Other: Respiratory and psychological rehabilitation — Respiratory rehabilitation consists of 12 sessions of respiratory and physical exercises that patients perform at home with the help of a physiotherapist. Sessions have 1 hour of duration and are performing twice a week. Exercises include (1) Training of the respiratory muscles through pursed-lip breaths. (2) Effective cough exercises. (3) Diaphragmatic contractions in a supine position with a lightweight placed on the anterior abdominal wall. (4) Stretching exercise of extremities and the back.
  The psychological support consists of 1 session to make the psychological history of the participant, and 6 sessions of emotion-centered problem-solving therapy, with cognitive-behavioral components and psychological management of emergencies and crises. These sessions have a 1-hour duration and are telephone-provided once a week by psychologists following the guidelines of the Inter-Agency Standing Committee on Mental Health and Psychosocial Support in Humanitarian and Disaster Emergencies.
  Arms: Home-based Respiratory Physiotherapy and Telephone-Based Psychological Support

SUMMARY:
Some COVID-19 survivors may have respiratory and mental health sequelae, especially those who required hospitalization. The investigators hypothesize that the participation of a rehabilitation program composite by home-based respiratory physiotherapy and telephone-based psychological support will improve respiratory function, quality of life, and psychological status in severe COVID-19 patients.

DETAILED DESCRIPTION:
In Peru, almost one million persons have survived COVID-19 and initial reports indicate that could exist long-term health damage. This study aims to assess the efficacy of a 6-week rehabilitation program following hospital discharge for patients who had severe COVID-19. The program includes 12 sessions of home-based respiratory therapy that the patient will carry out with a physiotherapist and 7 sessions of telephone-based psychological support bring by a psychologist.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Be discharged from hospitalization with a COVID-19 confirmed diagnosis
* Be able of understanding study procedures
* Be able to give informed consent
* Required oxygen flow greater than 6lt/min or through a high flow device at any time during hospitalization
* Have been evaluated by the rehabilitation service at least once during the hospitalization

Exclusion Criteria:

* Contraindications to six-minute walk test
* Contraindications to spirometry
* Complications during the baseline six-minute walk test
* Have neurological pathology, neuropathy, limb dysfunction, or other underlying physical disability that makes physical exercise impossible
* Be pregnant or breastfeeding
* Do not have access to the Internet or a telephone line
* Have previous lung diseases like asthma, COPD, fibrosis, or tuberculosis
* Moderate or severe heart disease (Grade III or IV, New York Heart Association)
* Have had another severe disease in the last six months
* Severe depression or suicidal intention
* Be taking any medication for depression, anxiety, or other medication prescribed by a psychiatrist prior to the onset of a COVID-19 condition
* Have cognitive impairment or sensory disturbance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Six minute walk distance | Change from baseline measure at hospital discharge to week 7 and 12
  Distance walked during 6-minutes (meters)

SECONDARY OUTCOMES:
Forced expiratory volume in the first second | Change from baseline measure at hospital discharge to week 7 and 12
  Measured in milliliters by dynamic spirometry
Forced Vital Capacity | Change from baseline measure at hospital discharge to week 7 and 12
  Measured in milliliters by dynamic spirometry
Quality of life assessed by the Short Form Health Survey (SF-36) questionnaire | Change from baseline measure at hospital discharge to week 7 and 12
  The SF-36 questionnaire consists of 36 items, which are used to calculate eight subscales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The first four scores can be summed to create the physical composite score (PCS), while the last four can be summed to create the mental composite score (MCS). Scores for the SF-36 scales range between 0 and 100, with higher scores indicating a better health-related quality of life
Quality of life assessed by the Health-Related Quality of Life (EQ-5D) questionnaire | Change from baseline measure at hospital discharge to week 7 and 12
  EQ-5D is a standardized tool for the assessment of quality of life in 5 different dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression). Possible scores range from 1 (No problem) to 3 (Extreme problems) and each dimension are evaluated individually.
Depressive symptomatology assessed by the Patient Health Questionnaire (PHQ-9) | Change from baseline measure at hospital discharge to week 7 and 12
  The Patient Health Questionnaire-9 (PHQ-9) consists of nine items covering the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria for major depression scored on a four-point 0 (not at all) to 3 (almost every day) scale, with total scores ranging from 0 to 27. A greater score means worse depressive symptoms.
Anxious symptoms assessed by the Generalized Anxiety Disorder (GAD-7) questionnaire | Change from baseline measure at hospital discharge to week 7 and 12
  The Generalized Anxiety Disorder-7 (GAD-7) consists of seven items covering the DSM-IV criteria for GAD scored on a four-point 0 (not at all) to 3 (almost every day) scale, with total scores ranging from 0 to 21. A higher score means worse anxiety symptoms.
Post-traumatic stress disorder symptomatology assessed by the Impact of Event Scale Revised (IES-R) questionnaire. | Change from baseline measure at hospital discharge to week 7 and 12
  IES-R consists of 21 items covering the DSM-IV criteria for PTSD. Score varying from 0 (no risk of post traumatic stress) to 88 (highest risk of post traumatic stress).
Impact on overall health by respiratory diseases assessed by the score of the St. George's respiratory questionnaire (SGRQ) | Change from baseline measure at hospital discharge to week 7 and 12
  The SGRQ scores from 0 (no impairment of quality of life by respiratory diseases/symptoms) to 100 (highest impairment of quality of life by respiratory diseases/symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Andres G Lescano, PhD, MHS, Principal Investigator — Universidad Peruana Cayetano Heredia; William Checkley, MD, PhD, Principal Investigator — Johns Hopkins University; Stella M Hartinger, MSc, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Hospital Nacional Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
Results will be published in an indexed peer-review journals.

REFERENCES:
- [Background] Spagnolo P, Balestro E, Aliberti S, Cocconcelli E, Biondini D, Casa GD, Sverzellati N, Maher TM. Pulmonary fibrosis secondary to COVID-19: a call to arms? Lancet Respir Med. 2020 Aug;8(8):750-752. doi: 10.1016/S2213-2600(20)30222-8. Epub 2020 May 15. No abstract available. PMID 32422177
- [Background] Xie L, Liu Y, Xiao Y, Tian Q, Fan B, Zhao H, Chen W. Follow-up study on pulmonary function and lung radiographic changes in rehabilitating severe acute respiratory syndrome patients after discharge. Chest. 2005 Jun;127(6):2119-24. doi: 10.1378/chest.127.6.2119. PMID 15947329
- [Background] Das KM, Lee EY, Singh R, Enani MA, Al Dossari K, Van Gorkom K, Larsson SG, Langer RD. Follow-up chest radiographic findings in patients with MERS-CoV after recovery. Indian J Radiol Imaging. 2017 Jul-Sep;27(3):342-349. doi: 10.4103/ijri.IJRI_469_16. PMID 29089687
- [Background] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Background] Yang LL, Yang T. Pulmonary rehabilitation for patients with coronavirus disease 2019 (COVID-19). Chronic Dis Transl Med. 2020 May 14;6(2):79-86. doi: 10.1016/j.cdtm.2020.05.002. eCollection 2020 Jun. PMID 32411496
- [Background] Liu K, Zhang W, Yang Y, Zhang J, Li Y, Chen Y. Respiratory rehabilitation in elderly patients with COVID-19: A randomized controlled study. Complement Ther Clin Pract. 2020 May;39:101166. doi: 10.1016/j.ctcp.2020.101166. Epub 2020 Apr 1. PMID 32379637
- [Background] Jang MH, Shin MJ, Shin YB. Pulmonary and Physical Rehabilitation in Critically Ill Patients. Acute Crit Care. 2019 Feb;34(1):1-13. doi: 10.4266/acc.2019.00444. Epub 2019 Feb 28. PMID 31723900
- [Derived] Soriano-Moreno AN, Flores EC, Hartinger SM, Mallma CY, Diaz AA, Gianella GE, Galvez-Buccollini JA, Coico-Lama AH, Malaga G, Fajardo E, Paredes-Angeles R, Otazu-Alfaro S, Lescano AG, Checkley W; WAYRA Trial Investigators. Home-Based Respiratory Physiotherapy and Telephone-Based Psychological Support for COVID-19 Survivors in Peru: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 24;11(10):e36001. doi: 10.2196/36001. PMID 36108135